CLINICAL TRIAL: NCT01561781
Title: A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Digoxin in Healthy Subjects When Administered Alone and in Combination With a Single Dose of Vandetanib (CAPRELSA) 300 mg
Brief Title: Study in Healthy Volunteers to Assess the Pharmacokinetics (PK) of Digoxin Administered Alone and in Combination With Vandetanib
Acronym: Vandetanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4200C00100
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; healthy volunteers; pharmacokinetics; vandetanib; digoxin
MeSH Terms: interventions — Digoxin; vandetanib

ARMS (1):
- digoxin then digoxin + vandetanib (Experimental): Digoxin alone followed by digoxin in combination with vandetanib
  Interventions: Drug: Digoxin; Drug: Vandetanib

INTERVENTIONS:
Drug: Digoxin — Oral tablets 0.25mg, single dose
Drug: Vandetanib — Oral tablets, 300 mg, single dose

SUMMARY:
This is a study in healthy volunteers to assess the pharmacokinetics (PK) of Digoxin administered alone and in combination with Vandetanib.

DETAILED DESCRIPTION:
A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of Digoxin in Healthy Subjects When Administered Alone and in Combination with a Single Dose of Vandetanib (CAPRELSA) 300 mg

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study
* specific procedures Volunteers must be males or females aged 18 to 45 years and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2,
* inclusive Females must have a negative pregnancy test at screening and on admission to the study center. Females must not be lactating and must be of non-childbearing potential defined as postmenopausal or documentation of irreversible surgical sterilization.

Exclusion Criteria:

* History of any clinically significant disease or disorder such as gastrointestinal, hepatic, renal or skin disease.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity,
* Volunteers who are current smokers and have smoked or used nicotine products within the previous 6 months
* Screening blood pressure of greater than 140/90 mmHg and/or a resting heart rate of less than 45 beats per minute (repeat test allowed at the Investigator's discretion
* Clinically significant abnormal12-lead ECG as assessed by the Investigator, QTcF interval greater than 450 ms
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV), or positive screen for drugs of abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
AUC for digoxin administered alone and in combination with vandetanib 300 mg | Predose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 18, 30, 48, 72, 96, 120, 144, and 168 hrs post dose
Cmax for digoxin administered alone and in combination with vandetanib 300 mg | Predose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 18, 30, 48, 72, 96, 120, 144, and 168 hrs post dose

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Treatment period + 7-14 days
ECG data | Treatment period + 7-14 days
Laboratory data | Treatment period + 7-14 days
Vital signs data | Treatment period + 7-14 days
Other PK parameters for digoxin administered alone and in combination with vandetanib 300 mg | Predose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, 12, 18, 30, 48, 72, 96, 120, 144, and 168 hrs post dose
Digoxin PK parameters for vandetanib in combination with digoxin | Predose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 48, 72, and 96 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Johansson S, Read J, Oliver S, Steinberg M, Li Y, Lisbon E, Mathews D, Leese PT, Martin P. Pharmacokinetic evaluations of the co-administrations of vandetanib and metformin, digoxin, midazolam, omeprazole or ranitidine. Clin Pharmacokinet. 2014 Sep;53(9):837-47. doi: 10.1007/s40262-014-0161-2. PMID 25117183
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1435&filename=CSR-D4200C00100.pdf
- See also: CSR-D4200C00100.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1435&filename=CSR-D4200C00100.pdf
- See also: Revised_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1435&filename=D4200C00100_Revised_CSP_redacted.pdf